CLINICAL TRIAL: NCT00501670
Title: A Non-therapeutic Study to Validate the Sampling Method to Confirm Presence of Varicella-zoster Virus (VZV) DNA by PCR in Clinical Samples From Lesions Collected From Adults (≥50 Years) With Clinically Diagnosed Herpes Zoster
Brief Title: VZV PCR Sampling Validation Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 109999
Record Dates: First submitted 2007-06-28; First posted 2007-07-16 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Herpes Zoster
Keywords: Herpes zoster; PCR; Varicella zoster Virus (VZV); Shingles; GSK Biologicals
MeSH Terms: conditions — Herpes Zoster; Chickenpox | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lesion samples

GROUPS / COHORTS (1):
- Group A: Collection of lesion samples and blood sampling from subjects aged >=50 years with clinically diagnosed herpes zoster
  Interventions: Procedure: Herpes zoster sampling procedure for VZV PCR; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Herpes zoster sampling procedure for VZV PCR — Four types of HZ lesions will be collected (Swabs of vesicles, Swabs of papules, Swabs of crusts and Crusts), 3 replicates of each.
Procedure: Blood sampling — Two blood samples taken, the first at the time of HZ diagnosis and the second one month later.

SUMMARY:
This study will evaluate and compare various methods for collecting lesion samples from subjects with clinically diagnosed herpes zoster for the laboratory confirmation of herpes zoster. The samples will be tested by polymerase chain reaction (PCR) to detect VZV DNA. Multiple samples from each type of herpes zoster lesion will be collected in order to determine whether the analysis of duplicate samples enhances the sensitivity of VZV DNA detection for the diagnosis of herpes zoster. In addition, blood will be collected for the evaluation of VZV immunity at the time of the initial herpes zoster sample collection (after herpes zoster has been clinically diagnosed) and one month later in order to establish the range of cellular and humoral immune responses during natural herpes zoster in adults ≥50 years old.

DETAILED DESCRIPTION:
This non-prophylactic, non-therapeutic study involves NO treatment of study participants.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with herpes zoster by the investigator including the presence of a typical herpes zoster rash.
* A male or female aged 50 years or older at the time of the subject's enrolment.
* Written informed consent obtained from the subject.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.

Exclusion Criteria:

* Any malignancy for which the subject is receiving active treatment, or any haematological malignancy.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within three months prior to the first vaccination, including corticosteroids, except inhaled and topical steroids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous vaccination against herpes zoster.
* Confirmed or suspected immunosuppression, based on medical history or physical examination (no laboratory testing required).
* A family history of congenital or hereditary immunodeficiency.
* History of or chronic alcohol or drug abuse.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: German male or female patients aged 50 years or older who are clinically diagnosed with HZ by the investigator including the presence of a typical HZ rash.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of VZV DNA copies per clinical sample collected. | At the time of the clinical diagnosis of HZ (Month 0).
Number of HSV DNA copies per clinical sample collected. | At the time of the clinical diagnosis of HZ (Month 0).
Number of actin DNA copies per clinical sample collected. | At the time of the clinical diagnosis of HZ (Month 0).

SECONDARY OUTCOMES:
Frequencies of CD4/CD8 T cells with antigen-specific IFN-g and/or IL-2 and/or TNF-α and/or CD40L secretion/expression to gE. | At Months 0 and 1.
Frequencies of CD4/CD8 T cells with antigen-specific IFN-g and/or IL-2 and/or TNF-α and/or CD40L secretion/expression to VZV. | At Months 0 and 1.
Anti-gE Ab concentrations. | At Months 0 and 1.
Anti-VZV Ab concentrations. | At Months 0 and 1.
Frequencies of gE-specific memory B cells. | At Months 0 and 1.
Frequencies of VZV-specific memory B cells. | At Months 0 and 1.
Occurrence of all SAEs. | During the whole study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (3):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Kiel, Schleswig-Holstein